CLINICAL TRIAL: NCT01897753
Title: Retrospective Study Of The Influence Of Age At Start Of Growth Hormone (Gh) Treatment On Height Gain In Children Born Small for Gestational Age (SGA)
Brief Title: Retrospective Study Of The Influence Of Age At Start Of Growth Hormone Treatment On Height Gain In Children Born Small for Gestational Age
Acronym: GH-RAST
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6281310
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Small For Gestational Age (SGA)
Keywords: SGA; Growth hormone
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Small For Gestational Age (SGA) Children: SGA children under growth hormone treatment for more than 36 months.
  Interventions: Drug: growth hormone

INTERVENTIONS:
Drug: growth hormone — 36 months

SUMMARY:
The purpose of this protocol is to retrospectively study the influence of age at start of growth hormone (GH) treatment on height gain in children born small for gestational age (SGA).

ELIGIBILITY:
Inclusion Criteria:

* SGA children.

  * Treated with GH at least 36 months.

Exclusion Criteria:

* Patients treated with GH for other indications (not SGA).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SGA children treated with GH at least 36 months
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
height SDS | 36 months
  height SDS of SGA children after 36 months of treatment

SECONDARY OUTCOMES:
height increase | 36 months
Change from Baseline in Lipid Parameters at Month X | 36 months
  Mean Total Cholesterol (TC), Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), and Triglyceride blood concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Spain (12):
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Capio H.Universitario Sagrat Cor, Barcelona, Barcelona
  - H. Vall d'Hebron, Barcelona, Barcelona
  - H. Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - H.Marqués de Valdecilla, Santander, Cantabria
  - H.Gregorio Marañón, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Virgen del Camino, Pamplona, Navarre
  - H.Clinico Universitario Valladolid, Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281310&StudyName=Retrospective%20Study%20Of%20The%20Influence%20Of%20Age%20At%20Start%20Of%20Growth%20Hormone%20Treatment%20On%20Height%20Gain%20In%20Children%20Born%20Small%20for%20Gestation